CLINICAL TRIAL: NCT00001162
Title: Study of Patients With Parasitic Infections of the Gastrointestinal Tract
Brief Title: Parasitic Infections of the Gastrointestinal Tract
Status: Terminated | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 770094; 77-I-0094
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-05-31

CONDITIONS: Amebiasis; Cryptosporidiosis; Giardiasis; Parasitic Disease; Parasitic Intestinal Disease; Gastrointestinal Helminth Infections
Keywords: Giardia; Helminth; Cryptosporidium; Hookworms; Trichuris; Strongyloides; Protozoa; Small Bowel Biopsy; E. Histolytica; Duodenal Aspiration; Coccidiosis; Clonorchis; Amebiasis; Parasitic Disease; Tapeworm; Trichinosis; Gastrointestinal Trematodes; Opisthorchis; Paragonimiasis; Echinococcus
MeSH Terms: conditions — Amebiasis; Cryptosporidiosis; Giardiasis; Parasitic Diseases; Intestinal Diseases, Parasitic; Hookworm Infections; Coccidiosis; Cestode Infections; Trichinellosis; Paragonimiasis; Echinococcosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
This protocol offers diagnosis and standard medical treatment for various parasitic gastrointestinal infections. Gastrointestinal parasites are either worms (helminths) or one-celled animals called protozoans which live in the human intestines. Often, parasitic infections do not cause illness. In these cases, drug treatment is not indicated, because treatment can have adverse side effects. Patients will be examined for their immune responses, correlation between the number of parasites and disease, and other studies.

Individuals with known or suspected parasitic diseases of the gastrointestinal tract, including amebiasis, giardiasis, hookworm, strongyloidiasis, trichuriasis, pinworm, tapeworm, trichinosis, clonorchis, opisthorchis, coccidiosis, paragonimiasis, and echinococcus may be eligible for this study.

Patient evaluations may include blood and urine tests, stool examination, X-rays, ultrasound studies and, uncommonly, duodenal aspiration for examination of fluid from the duodenum (first part of the small intestine). Other tests may be required, depending on the parasite and disease. Direct examination of the tissues of the intestines may be required to rule out certain infections.

Research procedures include collection of stool, blood and duodenal fluid when the diagnosis has been established and these procedures are not required for medical care. Patients with strongyloidiasis may also be given a diagnostic skin test similar to skin tests for tuberculosis and allergies. Research procedures on children will be limited to collection of stool, urine and blood. No more than 7 milliliters (1 1/2 teaspoons) per kilogram (2.2 pounds) body weight of blood will be collected in children over a 6-week period. In adults no more than 30 tablespoons of blood will be collected in a 6-week period.

Parasites may fail to respond to treatment. In these cases, it may be necessary to grow the parasite in the laboratory in order to test treatments in the test tube. Patients who do not respond to standard medications and dosing may need different doses of drugs or drugs or combinations of drugs used in the United States for other medical problems. If these medications or doses are used, patients will be informed of their possible side effects.

DETAILED DESCRIPTION:
The precis of this protocol is to allow the evaluation, treatment and study of patients with a variety of gastrointestinal parasites. This protocol primarily allows evaluation and treatment of patients with any intestinal parasite that requires a medical evaluation. The treatment and evaluation consists of standard of care. Research aspects include the collection and study of different parasite populations, analysis of the immune responses of the host, a correlation between parasite burden in the host and disease. These patients also serve as a source of reagents such as feces, white blood cells, and serum. The off-label use of FDA approved drugs is employed to treat symptomatic giardiasis in patients who cannot be cured otherwise and to determine empirically which regimens are effective and safe.

ELIGIBILITY:
* INCLUSION CRITERIA:

Persons with proven or highly suspected parasitic infections involving the gastrointestinal tract (including amebiasis, giardiasis, hookworm, strongyloidiasis, trichuriasis, pinworm, tapeworm, cyclorsporiasis, cryptosporidia infections, microsporidia infections, isosporidium infections, trichinosis, gastrointestinal dwelling trematodes, coccdioiosis, and echinococccus and additional infections).

Persons older than 2.

Ability and willingness of the subject or legal guardian/representative to give written informed consent.

EXCLUSION CRITERIA:

Subject unwilling or unable to comply with requirements of the protocol in the opinion of the investigator.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 1977-05-23; Study Completion 2017-05-31

PRIMARY OUTCOMES:
To Collect and study different parasite populations to study and/or axenization of specific parasites, analyze immune responses to homologous or heterologous parasites, and the development of diagnostic tests | Screening visit
Off label use of FDA approved drugs for treatment of Giardiasis in patients who cannot be cured otherwise, determining empirically which regimen is effective and safe | Post Tx follow up visit

CONTACTS AND LOCATIONS:
Overall Officials: Theodore E Nash, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kulakova L, Singer SM, Conrad J, Nash TE. Epigenetic mechanisms are involved in the control of Giardia lamblia antigenic variation. Mol Microbiol. 2006 Sep;61(6):1533-42. doi: 10.1111/j.1365-2958.2006.05345.x. PMID 16968226
- [Background] Ungar BL, Yolken RH, Nash TE, Quinn TC. Enzyme-linked immunosorbent assay for the detection of Giardia lamblia in fecal specimens. J Infect Dis. 1984 Jan;149(1):90-7. doi: 10.1093/infdis/149.1.90. PMID 6363569
- [Background] Nutman TB, Hussain R, Ottesen EA. IgE production in vitro by peripheral blood mononuclear cells of patients with parasitic helminth infections. Clin Exp Immunol. 1984 Oct;58(1):174-82. PMID 6478649